CLINICAL TRIAL: NCT05553899
Title: Utility of PET-MRI in Post-treatment Surveillance of Paediatric Brain Tumours: a Pilot Study
Brief Title: Utility of PET-MRI in Surveillance of Paediatric Brain Tumours
Acronym: PET-MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: GE Healthcare (Industry); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCH-2531
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2023-11

CONDITIONS: Brain Tumor, Pediatric
Keywords: Brain Tumor, children, PET, MRI
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (PET-MRI) (Experimental): Patients will undergo PET-MRI
  Interventions: Radiation: PET-MRI

INTERVENTIONS:
Radiation: PET-MRI — magnetic resonance imaging with positron emission tomography scanning using the tracer 18F-FDG

SUMMARY:
This is a pilot project to explore the utility of PET-MRI in the post-treatment surveillance of high-grade gliomas or medulloblastomas in children in our institution.

DETAILED DESCRIPTION:
Brain tumours are the most common solid tumours and the leading cause of death from cancer in children. A particular challenge in their management is detection of recurrent, residual or progressive tumour after initial treatment. This is typically detected on conventional MR surveillance scans. However, it is well documented that post-therapeutic changes can occur on MRI which may not represent disease, particularly after radiotherapy. Erroneously interpreting treatment-related changes as tumor progression may lead to the cessation of an effective treatment or the overestimation of the efficacy of a subsequent treatment. This is particularly important when assessing novel therapies in the context of early-phase clinical trials. A more accurate, non-invasive method of monitoring children after treatment for brain tumours could therefore enhance clinical management and may also lead to a more accurate assessment of novel therapies.

Hybrid Positron emission tomography-magnetic resonance imaging (PET/MRI) combines the high contrast and morphological resolution of MRI with the metabolic and physiological resolution from an intergrated PET scan. A variety of PET radiopharmaceutical tracers have been employed but 18F-fluodeoxyglucose (18F-FDG) has evolved over the last two decades to become the most important clinically. Increased glucose metabolism indicated by an increased FDG uptake is commonly seen in proliferating tumors due to the increased glucose transporter expression and the enzyme hexokinase, converting FDG to a phosphorylated product.

FDG-PET/CT has been demonstrated to have use for the differentiation of residual or recurrent tumours from post-therapeutic radiotherapy changes in adults 3-5 but its value in children is largely limited to case reports or small case series. The value of PET/MRI in paediatric in paediatric brain tumours is even less certain but in a series of 85 patients it was found to have a significant impact on management in the majority of cases. The accuracy of FDG PET in tumor surveillance may be higher than what has been historically reported because of improved spatial localization with concurrent use of MRI rather than CT.

This is a pilot project to explore the utility of PET-MRI in the post-treatment surveillance of high-grade gliomas or medulloblastomas in our institution. These tumours have the highest uptake of 18F-FDG and PET-MRI is therefore more likely to add diagnostic accuracy during their follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Have a presumptive or histologically confirmed diagnosis of a malignant brain tumour requiring treatment
* Diagnostic uncertainty about tumour recurrence post-treatment based on conventional MR imaging in the opinion of the MDT
* Have a life expectancy of at least three months
* Able to comply with an MRI scan without a general anaesthetic

Exclusion Criteria:

* Unable to comply with an MRI scan without a general anaesthetic
* Diabetes or other causes of hyperglycaemia
* Pregnancy
* Patient body habitus above scanner dimensions
* Standard contra-indication to MRI (eg. pacemaker, non-compatible metallic implants, altered renal function)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 1 year
  Explore whether it is possible to recruit and scan children for post-treatment surveillance of brain tumours using PET-MRI in Sheffield in our centre

SECONDARY OUTCOMES:
Acceptability | 1 year
  Are the study design, procedures, and intervention appropriate from the perspective of the participants?
Accuracy | 1 year
  determine the accuracy of FDG-PET vs MRI in determining residual tumour or tumour recurrence during post-treatment surveillance of high grade gliomas or medulloblastomas compared with biopsy results or clinical and radiological follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Rominyi, MBChB, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Children's Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No